CLINICAL TRIAL: NCT05848154
Title: A Single-center, Observational, Prospective Cohort Study of ctDNA Testing in Evaluation of Neoadjuvant Chemotherapy Efficacy and Exploration of Chemoresistance Mechanisms in Pancreatic Cancer
Brief Title: Application of ctDNA in Evaluation of Neoadjuvant Chemotherapy Efficacy and Exploration of Chemoresistance Mechanisms in Pancreatic Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Fudan University (Other); Amoy Diagnostics (Industry)
Responsible Party: Sponsor
Other Study IDs: ZSPAC-07
Record Dates: First submitted 2023-02-12; First posted 2023-05-08 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Patients With Non-metastatic Pancreatic Cancer; Evaluation of Tumor Resectability Shall be Made in Consensus at Multidisciplinary Meetings, According to NCCN Guideline Version 1.2022 Pancreatic Adenocarcinoma
Keywords: Pancreatic Neoplasms; Circulating tumor DNA; Neoadjuvant Therapy; Treatment Outcome
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ctDNA detection group: ctDNA detection, WES and RNA-seq will be performed on blood samples of all patients in this group.
  Interventions: Diagnostic Test: ctDNA detection

INTERVENTIONS:
Diagnostic Test: ctDNA detection — Blood samples are collected from patients at different time points during the monitoring process before treatment, after treatment, after surgery, and after adjuvant therapy/chemotherapy. ctDNA detection is performed on blood samples of all enrolled patients. WES and RNA-seq of samples from patients before and after treatment are performed to reveal the mechanisms of drug resistance.

SUMMARY:
The purpose of this study is to evaluate the value of ctDNA detection in the assessment of response rate to neoadjuvant chemotherapy in pancreatic cancer and to explore the correlation between ctDNA clearance and prognosis at different time points. Meanwhile, whole exome sequencing (WES) and RNA Sequencing (RNA-seq) of samples of responders and non-responders to neoadjuvant chemotherapy before and after treatment are performed to explore the mechanisms of drug resistance and provide guidance for clinical decision making.

DETAILED DESCRIPTION:
Pancreatic cancer is highly malignant with poor prognosis, and the overall 5-year survival rate is only about 9%. The value of neoadjuvant therapy in pancreatic cancer has been demonstrated by many studies, and a scientific and accurate evaluation of the efficacy of neoadjuvant therapy is crucial to its implementation and achieving the best outcomes. Circulating tumor DNA (ctDNA) analysis provides a non-invasive way to repeatedly assess the genomic profile of tumor. With improvements in detection techniques providing higher levels of sensitivity, ctDNA analysis is rapidly being accepted as a reliable tool in oncology. The purpose of this study is to evaluate the value of ctDNA detection in the assessment of response rate to neoadjuvant chemotherapy in pancreatic cancer and to explore the correlation between ctDNA clearance and prognosis at different time points. Meanwhile, whole exome sequencing (WES) and RNA Sequencing (RNA-seq) of samples of responders and non-responders to neoadjuvant chemotherapy before and after treatment are performed to explore the mechanisms of drug resistance and provide guidance for clinical decision making.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients with non-metastatic pancreatic cancer;
* The pathological features were identified as pancreatic ductal carcinoma;
* Patients with clinical risk factors including significantly elevated CA19-9 levels at diagnosis, large primary tumor volume, large regional lymph node diameter, significant weight loss, and extreme pain;
* Patients accept neoadjuvant chemotherapy voluntarily with the regimen of modified FOLFIRINOX, and disease evaluation should be conducted every two courses, surgery should be performed without delay if resection criteria have been met, and at least two courses of chemotherapy should be completed;
* Age ≥18 years old;
* No other tumor treatment within 4 weeks prior to enrollment;
* Complete clinical data, including basic information, pathological information, treatment information;
* The subjects voluntarily join the study and sign the informed consent with good compliance, and cooperate with the acquisition of tissue samples and regular blood samples.

Exclusion Criteria:

* Any other systemic antitumor therapy priorly;
* Concomitant malignancies under treatment;
* Patients with a history of allergy to relevant chemotherapy agents;
* Failure to comply with the requirements of the visit plan;
* Patients who may be absent from the visit period for 2 weeks or more during the treatment period;
* The researchers determine that the subjects have other factors that could have caused the study to be discontinued.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-metastatic pancreatic cancer. Evaluation of tumor resectability should be made in consensus at multidisciplinary meetings/discussions, according to NCCN guideline of pancreatic adenocarcinoma, Version 1.2022.
Sampling Method: Probability Sample
Enrollment: 92 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) of neoadjuvant therapy in patients with non-metastatic pancreatic cancer | Up to 24 months
  Pre-treatment ctDNA detection and mutation characterization in blood are used to evaluate objective response rate (ORR) of neoadjuvant therapy in patients with non-metastatic pancreatic cancer.

SECONDARY OUTCOMES:
Rate of adverse reactions | One week during therapy and 3 months thereafter up to 24 months.
  ctDNA detection is performed to evaluate the rate of adverse reactions to neoadjuvant therapy in patients with non-metastatic pancreatic cancer.
The correlation between detection of blood ctDNA and mutation characteristics before treatment and the rate of adverse reactions | One week during therapy and 3 months thereafter up to 24 months.
  ctDNA detection is performed to analyze the correlation between detection of blood ctDNA and mutation characteristics before treatment and the rate of adverse reactions.
The correlation between postoperative ctDNA in blood and clearance of ctDNA after adjuvant therapy and overall survival (OS) in patients with operable pancreatic cancer | One week during therapy and 3 months thereafter up to 48 months.
  Correlation between postoperative ctDNA in blood and clearance of ctDNA after adjuvant therapy and overall survival (OS) in patients with operable pancreatic cancer.
The recurrence of pancreatic cancer | One week during therapy and 3 months thereafter up to 24 months.
  Blood ctDNA after treatment is used to monitor the recurrence of pancreatic cancer.
The timeliness and accuracy of ctDNA with CA19-9 and medical imaging in the detection of disease recurrence | Up to 24 months.
  Blood ctDNA after treatment is used to compare the timeliness and accuracy of ctDNA with CA19-9 and medical imaging in the detection of disease recurrence.
The mechanisms of drug resistance to neoadjuvant chemotherapy | One week during therapy and 3 months thereafter up to 24 months.
  WES and RNA-seq of tissue samples of pancreatic cancer patients before and after treatment are performed to explore the mechanisms of drug resistance to neoadjuvant chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Wen-hui Wen-hui, MD, PhD, Principal Investigator — Shanghai Zhongshan Hospital; Wen-Quan Wang, MD, PhD, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
The IPD will not be shared with other researchers in order to protect patients' privacy.